CLINICAL TRIAL: NCT04181749
Title: Peri-vascular Adipose Tissue Inflammation Evaluated Using Coronary CT
Brief Title: Peri-vascular Adipose Tissue Inflammation Evaluated Using Coronary CT Angiography
Acronym: P-VECT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Collaborators: University of Oxford (Other); British Heart Foundation (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0719
Record Dates: First submitted 2019-11-19; First posted 2019-11-29 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — Aspirin; Atorvastatin

STUDY DESIGN:
Intervention Model Description: Patients randomized to No treatment or Aspirin and Statin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No treatment (No Intervention): Patients will not be prescribed aspirin and statin
- Aspirin and Atorvastatin (Active Comparator): Patients prescribed aspirin and atorvastatin
  Interventions: Drug: aspirin and atorvastatin

INTERVENTIONS:
Drug: aspirin and atorvastatin — Patients will be randomized and prescribed either no treatment or aspirin 75mg and Atorvastatin 40mg
  Arms: Aspirin and Atorvastatin

SUMMARY:
The P-VECT Study proposes to test the use of CCTA-derived FAI measurements in a group of patients with coronary artery inflammation, who will receive routinely-used statin and aspirin treatment. The P-VECT Study is a pilot study that will provide the rationale and data for power calculations to enable design of pivotal trials of the clinical effectiveness of FAI.

DETAILED DESCRIPTION:
In this research we will study the ability of coronary CT angiography (CCTA)- derived Fat Attenuation Index (FAI) measurements to detect changes in coronary artery inflammation following treatment with atorvastatin and aspirin . CT scan images are used to evaluate the presence of atherosclerotic plaque in the wall of the coronary arteries. The new CCTA technique, FAI, detects and quantifies coronary artery inflammation by analysis of the characteristics of the adipose tissue (fat) around the wall of the artery - the peri-vascular adipose tissue (PVAT) This is a pilot study, involving patients undergoing a clinically indicated CCTA as part of their routine clinical care who are shown (on their scans) to have mild coronary artery plaques (<50% luminal stenosis) with a high FAI value (>70.1 HU). Patients will have 6 visits (one of which screening) with hospital attendance on 3 occasions for blood tests and drug supply. The pilot study will provide the rationale for power calculations from which further studies can be developed to evaluate the clinical effectiveness of FAI.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following conditions:

1. Male or Female, aged 30 to 80 years,
2. CCTA scan showing mild coronary artery plaques (<50% luminal stenosis) with a high FAI value (>70.1 HU) within last 3 months.
3. No definite clinical indication for statin treatment (i.e. do not have either cholesterol >6.5 mM, or cholesterol >5.0 mM and QRISK score >10%).
4. Clinical equipoise for statin and aspirin treatment, as determined by the local treating physician. In these patients, there is clinical equipoise because routine treatment with aspirin and statin is not mandated by current guidelines, but the presence of minor coronary artery plaques is frequently interpreted by clinicians as an indication for aspirin and statin treatment. Accordingly, some patients in this group typically receive aspirin and statin treatment, whereas others do not.
5. Willing and able (in the Investigators opinion) to comply with all study requirements.
6. Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of any incidental findings.
7. Able to understand both verbal or written English

   -

Exclusion Criteria:

* The participant may not enter the study if ANY of the following are known to apply:

  1. Previous documented history of coronary artery disease requiring treatment. This includes any of the following:

     Acute myocardial infarction Unstable angina Coronary revascularization procedure Clinically significant coronary artery disease diagnosed by invasive or non-invasive testing.
  2. Known diabetes mellitus
  3. Definite clinical indication for statin treatment (i.e. has either cholesterol >6.5 mM, or cholesterol >5.0 mM and QRISK score >10%).
  4. Treatment with aspirin, statin or any prescribed lipid modification therapy in 6 weeks before baseline CCTA
  5. Atrial fibrillation (paroxysmal or persistent)
  6. History of New York Heart Association (NYHA) Class III or IV heart failure within the past 12 months of consent.
  7. Autoimmune disease requiring immunosuppressive therapy or systemic corticosteroid therapy
  8. Active treatment with any anti-inflammatory agents (e.g. NSAIDs, corticosteroids)
  9. Active neoplasm requiring surgery, chemotherapy, or radiation within the prior 12 months (subjects with a history of malignancy who have undergone curative resection or otherwise not requiring treatment for at least 12 months prior to screening with no detectable recurrence are allowed)
  10. Contraindication for aspirin and/or statin therapy
  11. Severe Chronic kidney disease (estimated glomerular filtration rate < 30 mL/min/1.73 m² and/or serum creatinine > 2.5 mg/dL or 220 µmol/l).
  12. Hepatic dysfunction (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] > 3 × the upper limit of normal [ULN] measured on local labs in last 6 months)
  13. Any clinically significant abnormality identified at the time of screening that, in the opinion of the Investigator, would preclude safe completion of the study.
  14. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
  15. Participants who have participated in another research study involving a treatment intervention or an investigational product, in the past 12 weeks.
  16. Patients unable to understand verbal or written English.
  17. Contraindication to contract dye for CCTA.
  18. Pregnancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate ability of new coronary CT angiogram (CCTA) scan biomarker- Fat Attenuation Index (FAI). | 3year study- Two years recruitment with 8 month patient follow up
  The overall objective is to evaluate the ability of a new cardiac CCTA scan technique, fat attenuation index (FAI), to detect changes in coronary artery perivascular fat inflammation following 8 months treatment with atorvastatin and aspirin medication

SECONDARY OUTCOMES:
Evaluate the association between changes in Fat Attenuation Index (FAI) and plasma lipid parameters. | 3year study- Two years recruitment with 8 month patient follow up
  Evaluate this association by measuring the % of change in plasma LDL-c.
Evaluate the association between changes in Fat Attenuation Index (FAI) and plasma lipid parameters. | 3year study- Two years recruitment with 8 month patient follow up
  Evaluate this association by measuring the % of change in plasma HDL-c.
Evaluate the association between changes in Fat Attenuation Index (FAI) and plasma lipid parameters. | 3year study- Two years recruitment with 8 month patient follow up
  Evaluate this association by measuring the % of change in triglycerides.
Evaluate the association between changes in FAI and plasma biomarkers of inflammation. | 3year study- Two years recruitment with 8 month patient follow up
  Evaluate this association by measuring the % of change in plasma IL-6.
Evaluate the association between changes in FAI and plasma biomarkers of inflammation. | 3year study- Two years recruitment with 8 month patient follow up
  Evaluate this association by measuring the % of change in plasma high sensitivity C-reactive protein (hsCRP) .

CONTACTS AND LOCATIONS:
Overall Officials: David Adlam, Dr., Principal Investigator — University Hospitals of Leicester and University of Leicester
Locations (3):
- United Kingdom (3):
  - University Hospitals of Leicester, Leicester
  - Royal Brompton Hospitals Trust, London
  - John Radcliffe Hospital, Oxford